CLINICAL TRIAL: NCT05100511
Title: Fundus Image-guided Focal Electroretinography, Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maculaser Oy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MACULARERG01
Record Dates: First submitted 2021-10-06; First posted 2021-10-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2021-11

CONDITIONS: Healthy; Macular Edema; Macular Degeneration
Keywords: Electroretinography; ERG
MeSH Terms: conditions — Macular Edema; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: The usability of the investigational device is examined first with 10 healthy subjects and afterwards with total of 10 patients suffering either from macular edema or macular degeneration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I, healthy subjects (Experimental): General usability of the device is tested with healthy patients. Different commercial electroretinography electrodes are tested to investigate the patient comfort, usability and signal-to-noise ratio when recording fundus image-guided focal electroretinography with the investigational device. Most suitable electrode is selected to phase II.
  Interventions: Device: ERG electrode tests for fundus image-guided focal ERG
- Phase II, patients with macular edema or macular degeneration (Experimental): The usability of the device is tested with patients suffering either from macular edema or macular degeneration. Fundus image-guided focal electroretinography is recorded with the electrode chosen in phase I from two different retinal areas: from an area with macular edema or signs of macular degeneration and from a healthy area (area without macular edema or signs of macular degeneration).
  Interventions: Device: Fundus image-guided focal ERG

INTERVENTIONS:
Device: ERG electrode tests for fundus image-guided focal ERG — Investigate the patient comfort, usability and signal-to-noise ratio of different commercial CE marked ERG electrodes.
  Arms: Phase I, healthy subjects
Device: Fundus image-guided focal ERG — Record focal ERG from a healthy retinal area and from an area with visible symptoms.
  Arms: Phase II, patients with macular edema or macular degeneration

SUMMARY:
The purpose of this study is to investigate the usability of fundus image-guided focal electroretinography device with healthy subjects and with macular edema and macular degeneration patients.

DETAILED DESCRIPTION:
In this study, we will study the usability of focal electroretinography device combined with slit lamp biomicroscope. The device allows simultaneous fundus imaging and focal ERG recording from the desired retinal area.

In phase I, the usability of the investigational device is tested with 10 healthy volunteers. The examinations include focal ERG and noise tests with commercial ERG electrodes. The stimulus lights are guided to the fundus using either non-contact of contact fundus lens. One electrode is selected for phase II based on signal-to-noise ration, usability, and comfort.

In phase II, fundus image-guided focal ERG recordings are conducted with total of 10 patients having either macular edema or macular degeneration. The aim of the phase II is to test whether the investigational device can be used to record focal ERG signal from the desired symptomatic retinal area.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with no signs of macular edema or macular degeneration (phase I)
* Patients with either macular edema or macular degeneration (phase II)
* Able to give informed consent

Exclusion Criteria:

* Epileptic patients
* Vulnerable population: pregnant and breastfeeding women, underage, prisoners, persons with physical handicaps or mental disabilities, and disadvantaged persons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Signal-to-noise ratio of focal electroretinography signal | Through study completion, an average of 1 year
  Signal-to-noise ratio of the focal ERG signals with different ERG electrodes.
Focal ERG from symptomatic retinal area | Through study completion, an average of 1 year
  Explore the device feasibility in recording focal ERG signal from areas with macular edema or macular degeneration.

SECONDARY OUTCOMES:
Patient comfort and usability of different ERG electrodes in focal ERG. | Through study completion, an average of 1 year
  Investigated using a questionnaire for the subjects and investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Joni Turunen, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Retinal Outpatient Clinic, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No